

Harvard University-Area
Committee on the Use of Human Subjects
44-R Brattle, Suite 200 (2nd floor)
Cambridge, MA 02138
IRB Registration - IRB00000109
Federal Wide Assurance - FWA00004837

## **Notification of Modification / Update Approval**

November 20, 2020

Peter Franz pfranz@g.harvard.edu

**Protocol Title:** Testing whether selected blog posts can improve well-being

Principal Investigator: Peter Franz
Protocol #: IRB19-0843
Submission #: MOD19-0843-02

Funding Source: Matt Nock's seed fund

Review Date: 11/20/2020
MOD Effective Date: 11/20/2020
IRB Review Type: Expedited
IRB Review Action: Approved

The Institutional Review Board (IRB) of the Harvard University-Area approved this Modification / Update.

The purpose of this study modification is to increase enrollment numbers, update compensation, and remove sharing of results with participants.

The documents that were finalized for this submission may be accessed through the IRB electronic submission management system at the following link: <a href="IRB19-0843">IRB19-0843</a>

The IRB made the following determinations:

• Risk Determination: No greater than minimal risk

While the below message may not be applicable to this study, we are including this message on all study actions so that the Harvard research community is aware of current guidance.

The resumption of in-person research will occur in phases with timing based on governmental policies and the state of the disease, the health care system, and society at large. The principal investigator (PI) of a research program/study will be required to craft a plan outlining the COVID-19 precautions that will be undertaken for their research. The researcher's plans will be subject to School/Departmental review and approval. No in-person research can begin until a researcher's plan receives School/Departmental approval.



Instructions on how to get approval for in-person research from your School/Department may be found here - <a href="https://cuhs.harvard.edu/instructions-returning-person-human-subjects-research?admin\_panel=1">https://cuhs.harvard.edu/instructions-returning-person-human-subjects-research?admin\_panel=1</a> You will also find on this site an outlined process, guidance, templates, and standard operating procedure examples to assist researchers and their Schools/Departments to get in-person human subjects research up and running.

## NOTE!

- ✓ Should a researcher receive approval from their School/Department for in-person human subjects research and their study is taking place at a location outside of Harvard, it is important that these studies follow any guidelines or instructions from the specific facility where in-person research would occur. As some research may occur in another state, with another institution, or under the direction of another IRB (as in a reliance agreement situation), this is especially important. It is the responsibility of the Study Team to keep apprised of potential restrictions and conduct their study accordingly.
- ✓ Harvard Affiliates should note any travel and other restrictions that are in place by visiting the Harvard COVID-19 website https://www.harvard.edu/coronavirus.

Please know that the default for all research involving in-person contact is to be paused. To the extent possible, study activities that can be done remotely by telephone or electronically, such as screening or follow-up, should be done in this way.

Should further restrictions pertaining to contact with study subjects be imposed at any time, it is the responsibility of the study team to follow guidance regarding when to pause a study and contact the HUA IRB.

Monitor the HUA IRB website < <a href="https://cuhs.harvard.edu/questions-about-covid-19-and-your-research">https://cuhs.harvard.edu/questions-about-covid-19-and-your-research</a> for updates.

Please contact me at 617-496-1185 or mikaela\_niemasz-cavanagh@harvard.edu with any questions.

Sincerely,

Mikaela Niemasz-Cavanagh IRB Administrator